CLINICAL TRIAL: NCT02613546
Title: THE INFLUENCE OF COGNITIVE BEHAVIORAL THERAPY IN SEXUAL DYSFUNCTION FEMALE: Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-11754978
Record Dates: First submitted 2015-11-22; First posted 2015-11-24 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Sexual Dysfunctions
Keywords: cognitive-behavioral psychotherapy; Sexual Dysfunctions; Women
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral therapy (CBT) (Experimental): The study group will undergo 10 sessions of guidelines and cognitive behavioral therapy (CBT) about an hour long, once a week. Of these:
  1. evaluation session;
  2. sessions of psychoeducation about the CBT model
  5 sessions of cognitive restructuring 2 sessions of preventing relapse
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- Control (Other): The control group will be subjected to 10 weekly sessions (1 time per week) approximately one hour guidelines.
  Interventions: Behavioral: Control therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — The study group will undergo 10 sessions of guidelines and cognitive behavioral therapy (CBT) about an hour long, once a week. Of these:
  1. evaluation session;
  2. sessions of psychoeducation about the CBT model
  5 sessions of cognitive restructuring 2 sessions of preventing relapse
  Arms: Cognitive behavioral therapy (CBT)
Behavioral: Control therapy — The control group will be subjected to 10 weekly sessions (1 time per week) approximately one hour guidelines.
  Arms: Control

SUMMARY:
This research is a randomized clinical trial aims to evaluate the influence of cognitive-behavioral psychotherapy (CBT) on quality of life and sexual function of patients with sexual dysfunction. The notion of sexual health for the World Health Organization exceeds the concept of sickness absence, having a subjective well-being of significance in the spheres of self-concept, self-image, interpersonal relationships and sense of self worth. Furthermore, sexual satisfaction and relationship quality of life is also evidenced in many studies. CBT is a brief and focal psychotherapy with proven efficacy in several mental disorders, improving health and quality of life of the treated populations. However, they did not find clinical trials that showed the effectiveness of CBT in Sexual Dysfunctions. This study aims to then fill this gap by evaluating the relationship from the use of techniques of CBT.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-59 years;
* FSFI less than or equal to 26.

Exclusion Criteria:

* Scores of Beck Scales - moderate or severe;
* Prescribing hormone therapy after starting the group.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2015-09-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Score Function Sexual | one week
  After cognitive behavioral therapy will be held the FSFI questionnaire to assess whether there was change in the score and its domains.

SECONDARY OUTCOMES:
Quality of Life Scale Questionary | one week
  After cognitive behavioral therapy will be held the SF-36 questionnaire in which assesses the overall quality of life of women. The higher the score the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia V Lordelo, PhD, Principal Investigator — Centro de Atenção ao Assoalho Pélvico - BAHIANA
Locations (1):
- Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia, Brazil